CLINICAL TRIAL: NCT01972490
Title: Study of Avastin in Combination With Chemotherapy for the First Line Treatment of RAS Mutant Unresectable Colorectal Liver-limited Metastases
Brief Title: Avastin in Combination With Chemotherapy for RAS Mutant Unresectable Colorectal Liver-limited Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Jianmin Xu, PhD Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCMCLM
Record Dates: First submitted 2013-09-23; First posted 2013-10-30 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal neoplasms; liver metastasis; chemotherapy; avastin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Experimental): patients received avastin in combination with mFOLFOX6
  Interventions: Drug: avastin; Drug: mFOLFOX6
- ARM B (Active Comparator): Patients received mFOLFOX6 alone
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: avastin — Drug: avastin On day 1 of a 14 day treatment cycle, patients received a 2-hour infusion of avastin (5mg/kg) followed by chemotherapy of mFOLFOX6 until progressive disease or unacceptable toxicity.
  Other Names: Bevacizumab
  Arms: ARM A
Drug: mFOLFOX6 — mFOLFOX-6 (oxaliplatin, 85mg/m2 on day 1 infused during 2 hours;LV400mg/m2 on days 1 infused during 2 hours, followed by FU 400 mg/m2 intravenous bolus then 2400 mg/m2 continuous infusion for 46 hours)

SUMMARY:
In this study, the investigators assessed the effect of avastin in combination with chemotherapy in the treatment of RAS mutant-type, unresectable colorectal liver-limited metastases

DETAILED DESCRIPTION:
Patients will be eligible for inclusion if the patients have histologically confirmed colorectal adenocarcinoma with RAS mutant liver-confined metastases deemed non-resectable. Eligible patients will be randomly assigned to chemotherapy plus avastin (arm A) or chemotherapy alone (arm B). Treatment will continue until tumor response indicates suitability for surgery for liver metastases or until disease progression or unacceptable toxic effects. The primary endpoint is the conversion rate to radical resection for liver metastases，which will be assessed by local multidisciplinary team (includes more than three liver surgeons and one radiologist) with the use of contrast-enhanced CT or MRI after 4 cycles and then every other 4 cycles up to 12 cycles. To provide an objective assessment of changes in resectability, radiological images will be presented by a radiologist to more than 3 liver surgeons, who are blinded to the clinical data. Patients will be considered resectable if 50% or more of surgeons vote for radical resection of LM. For patients whose liver-metastases are assessed resectable, resection should be scheduled to be performed within 2~3 weeks of the last treatment cycle. Following resection, patients will be advised to continue the same therapeutic regimen until the treatments reach a sum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumour was histologically confirmed colorectal adenocarcinoma;
3. Together with clinical or radiological evidence of first occurrence of non-resectable liver-only metastases
4. With evidence of tumor RAS gene mutant status;
5. With at least one measurable tumor.
6. Performance status (ECOG) 0~1
7. A life expectancy of ≥ 3 months
8. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization)
9. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either AST or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
10. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Previous exposure to target therapy, chemotherapy, radiotherapy or intervention therapy for colorectal liver metastases.
2. Known or suspected extrahepatic metastases.
3. Patients with known hypersensitivity reactions to any of the components of the study treatments.
4. Having previously participated in a study which included a possibility of being allocated to avastin therapy (whether or not the patient actually received avastin)
5. Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or left ventricular ejection fraction (LVEF) below the institutional range of normal
6. Acute or sub-acute intestinal occlusion
7. Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
8. Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
9. Known drug abuse/ alcohol abuse
10. Legal incapacity or limited legal capacity
11. Pre-existing peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
the rate of patients converted to resection for liver metastases | 3 years
  To explore whether avastin in combination with chemotherapy as treatment could improve the resection rate in patients with RAS mutant-type, unresectable colorectal liver-limited metastases compared with chemotherapy alone.

SECONDARY OUTCOMES:
progression free survival | 3 years
  PFS will be defined as the period from the first day of avastin treatment or chemotherapy to the date of disease progression (PD) or to death. Patients without PD who discontinued the study for any reason is censored at the last on-study tumor assessment date.or distant(i.e. metastasis) disease recurrence or death.
overall survival | 3 years
  OS will be calculated from randomization to death from any cause or the date of the last follow-up, at which point the data will be censored.
tumor response | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Tang W, Ren L, Liu T, Ye Q, Wei Y, He G, Lin Q, Wang X, Wang M, Liang F, Cui Y, Xu J. Bevacizumab Plus mFOLFOX6 Versus mFOLFOX6 Alone as First-Line Treatment for RAS Mutant Unresectable Colorectal Liver-Limited Metastases: The BECOME Randomized Controlled Trial. J Clin Oncol. 2020 Sep 20;38(27):3175-3184. doi: 10.1200/JCO.20.00174. Epub 2020 Aug 4. PMID 32749938